CLINICAL TRIAL: NCT04629833
Title: A Randomised, Open-label, Multicentre, Phase 3 Trial of First-line Treatment With Mesenchymal Stromal Cells MC0518 Versus Best Available Therapy in Adult and Adolescent Subjects With Steroid-refractory Acute Graft-versus-host Disease After Allogeneic Haematopoietic Stem Cell Transplantation (IDUNN Trial)
Brief Title: Treatment Of Steroid-Refractory Acute Graft-versus-host Disease With Mesenchymal Stromal Cells Versus Best Available Therapy
Acronym: IDUNN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: medac GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC-MSC.1/aGvHD
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Steroid-refractory Acute Graft-versus-host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MC0518 (Experimental): Participants will receive MC0518 1-2 million cells/ kilogram infusions (based on body weight at the Screening Visit) once a week for 4 weeks (Visit Day 1, 8, 15, and 22). Participants with partial response (PR) on Day 28 will have 2 additional MC0518 infusions administered on Day 29 and 36.
  Interventions: Biological: MC0518
- Best Available Therapy (BAT) (Active Comparator): Participants will receive any one of the following systemic BATs based on the Investigator's decision: mycophenolate mofetil (MMF), extracorporeal photopheresis (ECP), anti-thymocyte globulin (ATG), everolimus, and ruxolitinib (RUX).
  Interventions: Biological: BAT

INTERVENTIONS:
Biological: MC0518 — MC0518 will be intravenously infused immediately after thawing.
  Arms: MC0518
Biological: BAT — BAT including MMF, ECP, ATG, everolimus, and RUX will be administered based on Investigator's decision.
  Arms: Best Available Therapy (BAT)

SUMMARY:
The primary purpose of this trial is to demonstrate the superiority of MC0518 compared to the first used best available therapy (BAT) with respect to overall response rate (ORR) at Day 28 and/or overall survival (OS) until Visit Month 24 in adult and adolescent subjects with steroid-refractory acute graft-versus-host disease (SR-aGvHD).

ELIGIBILITY:
Inclusion Criteria:

* Participant had a previous allogeneic HSCT as indicated for non-malignant (including inborn errors of metabolism, primary immunodeficiencies, haemoglobinopathies, and bone marrow failure syndromes) or haematological malignant disease, irrespective of human leukocyte antigen match
* Participant has been clinically diagnosed with Grade II to IV aGvHD at the Screening Visit
* Participant has experienced failure of previous first-line aGvHD treatment (ie, SR-aGvHD), defined as: a) aGvHD progression within 3 to 5 days of therapy onset with >= 2 mg/kg/day of prednisone equivalent or b) failure to improve within 5 to 7 days of treatment initiation with >= 2 mg/kg/day of prednisone equivalent or c) incomplete response after > 28 days of immunosuppressive treatment including at least 5 days with >= 2 mg/kg/day of prednisone equivalent
* Participant has an estimated life expectancy > 28 days at the Screening Visit
* Male or female participant who is >= 12 years of age at the Screening Visit

Exclusion Criteria:

* Participant has overt relapse or progression or persistence of the underlying disease at the Screening Visit
* Participant has received the last HSCT for a solid tumour disease
* Participant has GvHD overlap syndrome at the Screening Visit
* Participant has received systemic first line treatment for aGvHD other than steroids and a prophylaxis with other than calcineurin inhibitors, mammalian target of rapamycin (mTOR) inhibitors, anti-thymocyte globulin (ATG), mycophenolate mofetil (MMF), methotrexate (MTX), and / or cyclophosphamide before the Screening Visit
* Participant has a known pregnancy (as confirmed by a positive pregnancy test at the Screening Visit) and or is breastfeeding at the Screening Visit
* Participant has received treatment with any other investigational agent within 30 days or 5 half-lives (whichever is longer) before the Screening Visit (compliance to be confirmed for the period between the Screening Visit and the Baseline Visit at the Baseline Visit).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Overall Response (OR) | Day 28
  OR is defined as complete response (CR) or partial response (PR) at Day 28 relative to aGvHD status at baseline. CR is defined as resolution of aGvHD in all involved organs. PR is defined as improvement in 1 stage in 1 or more organs involved with aGvHD symptoms without progression in others. Number of participants with OR will be reported.
Overall Survival | Up to Month 24
  Overall survival is defined as the time from randomization to the date of death due to any cause.

SECONDARY OUTCOMES:
Freedom from Treatment Failure (FFTF) | Up to 6 months
  FFTF is defined as death, relapse or progression of the underlying disease, or addition or change to any further systemic immunosuppressive aGvHD therapy. Number of participants with FFTF will be reported.
Acute Graft-versus-host Disease (aGvHD) Response | Days 28, 60, 100 and 180
  Number of participants with aGvHD response will be reported. aGvHD response will be categorized as OR (CR + PR), CR, PR, and NR. NR is defined as the absence of CR or PR.
Change from Baseline in aGvHD Grades | Baseline and Days 8, 15, 22, 28, 60, 100 and 180
  aGvHD grades: Grade 0- no organ involvement (ie, Stage 0 skin, Stage 0 liver, and Stage 0 GI); Grade I-Stage 1 - 2 skin without liver/GI involvement; Grade II- Stage 3 skin and / or Stage 1 liver and / or Stage 1 GI; Grade III- Stage 2 - 3 liver and / or Stage 2 - 3 GI; Grade IV- Stage 4 skin and / or Stage 4 liver and/or Stage 4 GI.
Time to Response | Up to Month 24
  Time to response is defined as the time from the date of the first treatment administration to the date of response.
Duration of Response | Up to Month 24
  Duration is calculated from time from the first OR (CR or PR) until the time point of no aGvHD response in comparison to baseline.
Best Overall Response (OR) | Up to Day 28
  Best OR is defined as the achievement of an OR at any time point up to and including Day 28. Number of participants with best OR will be reported.
Cumulative Dose of Steroids for SR-aGvHD per Kilogram (kg) of Body Weight | Up to Day 60 and Month 24
  The cumulative dose of steroids given for SR-aGvHD per kg of body weight from baseline until Day 60 and until Visit Month 24 will be analyzed.
Number of Participants with Chronic Graft-versus-host Disease (cGvHD) | Day 60 to Month 24
  Number of participants with cGvHD will be reported.
Time to Chronic Graft-versus-host Disease (cGvHD) | Day 60 to Month 24
  Time to cGvHD is defined as the time between the last day of haematopoietic stem cell transplantation (HSCT) to the first episode of cGvHD.
Number of Participants with Graft Failure (GF) | Up to Month 24
  Number of participants with GF will be reported.
Number of Participants with Relapse or Progression in Participants with Underlying Malignant Disease | Up to Month 24
  Number of participants with relapse or progression in participants with underlying malignant disease will be reported.
Time to Relapse or Progression in Participants with Underlying Malignant Disease | Up to Month 24
  Time to relapse or progression in participants with underlying malignant disease will be reported.
Event-free survival (EFS) | Up to Month 24
  EFS is defined as the time from the date of randomization to the date of the event. An event is defined as GF, relapse or progression of the underlying disease, or death due to any cause.
Non-relapse Mortality (NRM) | Up to Month 24
  NRM is defined as the time from the date of randomisation to the date of the event. An event is defined as death without previous relapse or progression of the underlying disease.
Number of Participants with Adverse Events (AEs) and Adverse Reactions (ARs) | Until Day 60 or until 30 days after last administration of trial treatment, whichever is later (Up to Month 24)
Number of Participants with Adverse Events (AEs) and Adverse Reactions (ARs) by Severity | Until Day 60 or until 30 days after last administration of trial treatment, whichever is later (Up to Month 24)
  Severity will be graded based on Common Terminology Criteria for Adverse Events (CTCAE) v5.0: Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe; Grade 4- Life-threatening consequences; urgent intervention indicated; Grade 4- Death related to the AE.
Change from Baseline in Performance score based on Karnofsky scale (recipient age >= 16 years) | Baseline, Days 8, 15, 22, 28, 60 and 100
  The Karnofsky performance score (KPS), which is reported on an ordinal scale from 0 to 100, provides a rough measure of the participant's well-being, including their ability to conduct activities of daily living and functional capacity. Higher score indicates normal, no complaints and no evidence of disease.
Change from Baseline in Performance score based on Lansky Scale | Baseline, Days 8, 15, 22, 28, 60 and 100
  A Lansky score (recipient age greater than or equal to [>=] 1 years and less than [<] 16 years) will be recorded pre-treatment and measured serially at regular intervals after treatment. The score is a standard performance score that measures overall function of the child with a scale range from 0 to 100. Higher score indicates full activeness.
Change from Baseline in EuroQol-5D-5L (EQ-5D-5L): Health Status Index (HSI) | Baseline, Days 28, 60, 100 and 180
  EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ VAS. EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "TODAY". Responses were used to generate a HSI. HSI ranges from 0 (dead) to 1.00 (full health).
Change from Baseline in EuroQol-5D-5L (EQ-5D-5L): Visual Analogue Scale (VAS) | Baseline, Days 28, 60, 100 and 180
  EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ VAS. The EQ VAS self-rating records the respondent's own assessment of his or her overall health status at the time of completion, on a scale of 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Change from Baseline in Functional Assessment of Cancer Therapy-Bone Marrow Transplantation (FACT-BMT) Score | Baseline, Days 28, 60, 100 and 180
  The FACT-BMT questionnaire was designed to measure the quality of life in subjects undergoing bone marrow (BM) transplantation. It consists of the following categories of assessment: physical well-being, social / family well-being, emotional well-being, functional well-being, and additional miscellaneous concerns that the subject may have concerning their healthcare, persons involved in their life, and other emotions and incapabilities. Score ranges from 0-164, with higher score indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Kristin Möller, Study Director — medac GmbH
Locations (42):
- France (9):
  - Centre Hospitalier Universitaire (CHU) Amiens-Picardie - Hopital Sud, Amiens
  - CHU Jean Minjoz, Besançon
  - Hopital Michallon, Grenoble
  - CHRU Lille- Hopital Claude Huriez, Lille
  - CHU de Nantes - Hotel Dieu, Nantes
  - CHU de Nice Hopital Archet 1, Nice
  - Centre Hospitalier Lyon Sud Pavillon Marcel Berard 1G, Pierre-Bénite
  - Centre Hospitalier Universitaire CHU de Toulouse, Toulouse
  - Hopitaux De Brabois, Vandœuvre-lès-Nancy
- Germany (22):
  - Klinikum rechts der Isar, Munich, Bavaria
  - Universitaetsklinikum Wuerzburg - Medizinische Klinik und Poliklinik II - Zentrum fuer Allogene Blutstammzelltransplantation, Würzburg, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universitaet - Frankfurt am Main, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Uniklinik Koeln, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Essen - Klinik fuer Knochenmarktransplantation (KMT), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Universitaetsklinikum Leipzig, Selbststaendige Abteilung fur Haematologie und Internistische Onkologie, Leipzig, Saxony
  - Universitaetsklinikum Jena Klinik fuer Innere Medizin II, Haematologie und Onkologie, Jena, Thuringia
  - Universitaetsklinikum Jena - Klinik fuer Paediatrische Haematologie und Onkologie, Jena, Thuringia
  - Charite Universitaetsmedizin, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - University Hospital Bonn, Medizinische Klinik III, Bonn
  - Universitaetsklinikum Essen - Klinik fuer Paediatrische Haematologie und Onkologie, Essen
  - Klinikum der Johann Wolfgang Goethe University - University - Klinik fuer Paediatrische Haematologie und Onkologie, Frankfurt
  - Universitaetsklinikum Freiburg - Zentrum fuer Kinder- und Jugendmedizin (ZKJ) - Klinik fuer Paediatrische Haematologie und Onkologie, Freiburg im Breisgau
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitatsklinikum, Kiel
  - University Medical Center Mainz, Mainz
  - Universitaetsklinikum Mannheim, Mannheim
  - University Hospital Tuebingen Medical Center, Tübingen
- Poland (2):
  - Department of Pediatric Hematology, Oncology and BMT, Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie, Paastwowy Instytut Badawczy, Gliwice
- Spain (8):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario Vall dHebron, Barcelona
  - Institut Catal dOncologia, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Puerta De Hierro, Madrid
  - Hospital Universitario Carlos Haya, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i politecnic La Fe, Valencia
- Center for Allogeneic Stem Cell Transplantation and Cell Therapy (CAST), Karolinska Universitetssjukhuset Huddinge, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No